CLINICAL TRIAL: NCT03810612
Title: Continuity of Care, Adherence to Treatment and Self-reported Health After Percutaneous Coronary Intervention (CONCARD): a Patient-centered Care Study
Brief Title: Patient-reported Outcomes After Percutaneous Coronary Intervention
Acronym: CONCARD
Status: Active, not recruiting | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Stavanger HF (Other Government); Oslo University Hospital (Other); Zealand University Hospital (Other); Odense University Hospital (Other); Rigshospitalet, Denmark (Other); Herlev and Gentofte Hospital (Other); Western Norway University of Applied Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/57
Record Dates: First submitted 2018-12-21; First posted 2019-01-18 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease
Keywords: Adherence to treatment; Continuity of care; Health literacy; Patient involvement; Patient preferences; Percutaneous coronary intervention; Rehabilitation
MeSH Terms: conditions — Coronary Artery Disease; Treatment Adherence and Compliance; Patient Participation; Patient Preference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective is to investigate i) continuity of care, ii) health literacy and self-management, iii) adherence to treatment, and iv) patient preferences, healthcare utilization and costs, and to determine associations with future short- and long-term health outcomes in patients after percutaneous coronary intervention.

DETAILED DESCRIPTION:
CONCARD will use multiple designs. (1) An inductive exploratory design including in-depth interviews on patients' experiences of healthcare delivery will provide a context for the quantitative data to develop the content of the cohort study and trial intervention. (2) A prospective cohort design with a 1-year follow-up period will include data on patient-reported outcomes, and a 10-year follow-up for adverse events. In translation and adaptation of patient-reported outcome measures, a methodological design will be applied. (3) A discrete choice experiment will investigate patient preferences for aftercare and cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing percutaneous coronary intervention
* ≥ 18 years of age
* Living at home at the time of inclusion.

Exclusion Criteria:

* Patients who do not speak Norwegian/Danish
* Patients who are unable to fill in the questionnaires due to reduced capacities
* Institutionalized patients
* Patients with expected lifetime less than one year
* Percutaneous coronary intervention without stent implantation
* Patients undergoing percutaneous coronary intervention related to Transcatheter Aortic Valve Implantation or Mitraclip examination
* Previous enrollment in CONCARD (readmissions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone percutaneous coronary intervention will be included prospectively at each percutaneous coronary intervention centre.
Sampling Method: Non-Probability Sample
Enrollment: 3417 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Continuity of care | 2 months
  The Heart Continuity of Care Questionnaire (HCCQ) comprises 33 items covering eight topic areas regarding continuity of care. Respondents rate each item on a 6-point scale ranging from 1 (strongly disagree) to 5 (strongly agree) or 6 (not applicable).
Evaluation of the quality of healthcare delivery | 2 months
  The Nordic Patient Experiences Questionnaire (NORPEQ) comprises 8 items and gives a brief measure of patient experiences in evaluation of the quality of healthcare delivery. Respondents rate each item on a 5-point scale ranging from 1 (not at all) to 5 (to a large extent). Six of the eight NORPEQ items sum to produce an overall scale from 0 to 100, where 100 is the best possible experience of care.
Change in eHealth literacy | 2 months, 12 months
  The eHealth Literacy Scale (Eheals) is an 8-item measure of eHealth literacy developed to measure consumers' combined knowledge, comfort, and perceived skills at finding, evaluating, and applying electronic health information to health problems. Respondents indicate their agreement with statements on a 5-point Likert scale ranging from 1 (Strongly Disagree) to 5 (Strongly agree).
Change in health literacy | 2 months, 12 months
  The Health literacy questionnaire (HLQ) has nine scale scores that each measure an aspect of the multidimensional construct of health literacy. Each score provides insight into the strengths and limitations of the respondent, but the scores are most powerful when viewed together to show the 'health literacy profile' of the respondent.
Patient knowledge, skill, and confidence for self-management. | 6 months
  The Patient Activation Measure (PAM-13) comprises 13 items assessing patient knowledge, skill and confidence for self-management. Respondents indicate their agreement with statements on a 5-point Likert scale ranging from 1 (Strongly Disagree) to 4 (Strongly agree), or 5 (not applicable). Patients with a high activation score were associated with fewer mental health symptoms, greater recovery attitudes and medication adherence.
Change in beliefs and perceptions about medicines and treatment | 2 months, 6 months, 12 months
  The Beliefs about Medicines Questionnaire (BMQ) assesses beliefs and perceptions about medicines and treatment. The BMQ comprises two sections: the BMQ-Specific which assesses representations of medication prescribed for personal use and the BMQ-General which assesses beliefs about medicines in general. The two sections of the BMQ can be used in combination or separately. For this study, the BMQ-Specific will be used. Respondents rate 11 items on a 5-point scale ranging from 1 (strongly agree) to 5 (strongly disagree).
Change in self-reported adherence to medicines | 2 months, 6 months, 12 months
  The Medication Adherence Report Scale (MARS-5) measures self-reported adherence to medicines, it assesses both intentional and unintentional non-adherence. Respondents indicate their agreement with statements about their medicine use on a 5 point Likert scale ranging from 1 (always) to 5 (never).
Change in medication use | 2 months, 6 months, 12 months
  Data related to consumption of prescribed medication are identified through national prescription registries. The registries cover all prescriptions dispensed at pharmacies nationwide. The registries also include information about date of dispensation, quantity and strength dispensed. This will serve as complimentary information to patients' self-reported adherence.
Health care utilization | Up to 24 months
  Healthcare utilization will be assessed during follow-up, including patients' use of primary care services (general practitioner visits) and secondary care services (inpatient admissions and outpatient visits). The data source will be nationwide registries. The measurement unit will be mean number of visits.
Health care (associated) costs | Up to 24 months
  Health care (associated) costs will be valued using the tariffs of national agreements between the professional associations of medical specialists and the National Health Services. In secondary care, inpatient admissions and outpatient visits will be valued using the tariffs of the national case-mix system of the diagnosis-related groupings (DRG) and the ambulatory grouping system (DAGS). In addition, data will be collected on prescription of medication, which will be valued using the retail price. The data source will be nationwide registries. The measurement unit will be mean costs in Euros.

SECONDARY OUTCOMES:
Time to readmission to hospital | 30-days, 3 months, 6 months, 12 months, up to 10 years
  Cardiac and all cause readmissions
Time to death | 30-days, 3 months, 6 months, 12 months, up to 10 years
  Cardiac and all cause mortality
Change in anxiety and depression | 2 months, 6 months, 12 months
  The Hospital Anxiety and Depression Scale (HADS). The HADS is a fourteen item scale where seven of the items relate to anxiety and seven relate to depression. The respondent rates each item on a 4-point scale ranging from 0 (absence) to 3 (extreme presence). The total score is 42 (21 per subscale).
Change in self-reported health | 2 months, 6 months, 12 months
  EQ-5D-5L is an 5 item (plus a VAS scale) self-report-questionnaire assessing self-reported health. Each question has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Change in chest pain | 2 months, 6 months, 12 months
  The Seattle Angina Questionnaire (SAQ-7) comprises 7 dimensions of coronary artery disease. Each scale is transformed to a score of 0 to 100, where higher scores indicate better function (eg, less physical limitation, less angina, and better quality of life).
Change in fatigue | 2 months, 6 months,12 months
  A visual analog scale ranging from 0 (fatigue is not a problem) to 10 (fatigue is a major problem) is used to measure change in fatigue
Frailty status | 12 months
  The Study of Osteoporotic Fractures (SOF) index will be used to measure frailty status. The SOF index includes three items: 1) weight loss > 5% in the last year, 2) inability to rise from a chair five times without using arms, and 3) reduced energy level. The questions have dichotomous response alternatives (yes/no). Patients who meet none of these criteria will be considered robust, one of the criteria are pre-frail, and two or three of these criteria are considered frail.
Patient preferences in discrete choice experiments | 3 months
  A discrete choice experiment (DCE) is a quantitative technique for eliciting preferences to be used in the absence of revealed preference data. This involves asking individuals to state their preference over hypothetical alternative scenarios. Each alternative is described by several attributes which are used to determine if preferences are significantly influenced by these. No standardized measurement tool is used in DCE. The alternative scenarios (attributes) are developed for each individual study. Therefore, a DCE will be undertaken as a cross-sectional survey to investigate the preferences for aftercare. Participants are asked to choose between hypothetical aftercare programs described by five key characteristics that varies across each of the respondents' choices. The DCE will be carried out according to recommendations by the ISPOR group. A multinomial mixed logit model are used to model preferences and calculate marginal rates of substitution.
Health related quality of life | 12 months
  The HeartQoL questionnaire is a core ischemic heart disease specific health related quality of life (HRQL) questionnaire. The questionnaire comprises 14-items with 10-item physical and 4-item emotional subscales which are scored from 0 (poor HRQL) to 3 (better HRQL) with a global score if needed.
Change in physical and mental dimensions of health. | 2 months, 6 months, 12 months
  RAND-12 measures physical and mental dimensions of health. The 12 items in the questionnaire correspond to eight principal physical and mental health domains. The 12 items are summarized into two scores, a "Physical Health Summary Measure {PCS-physical component score}" and a "Mental Health Summary Measure {MCS-mental component score}".
Change in health status following myocardial infarction | 2 months, 6 months, 12 months
  The Myocardial Infarction Dimensional Assessment Scale (MIDAS) is a PRO measure developed and validated to specifically measure the health status of individuals who have suffered a myocardial infarction. It consist of 7 domains, and is a 35 item scale where respondents rate each item on a 5-point scale ranging from 1 (never) to 5 (always). The function of the MIDAS is to indicate the extent of ill health in each of the seven domains assessed, therefore each dimension is scored separately using a simple scoring methodology.

CONTACTS AND LOCATIONS:
Overall Officials: Tone M Norekvål, PhD, Principal Investigator — Haukeland University Hospital
Locations (7):
- Denmark (4):
  - Herlev and Gentofte Hospital, Copenhagen
  - Rigshospitalet, Copenhagen, Copenhagen
  - Odense University Hospital, Odense
  - Zealand University Hospital, Roskilde
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Rikshospitalet, Oslo
  - Stavanger University Hospital, Stavanger

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Norekval TM, Iversen MM, Oterhals K, Allore H, Borregaard B, Pettersen TR, Thompson DR, Zwisler AD, Breivik K. Perfect health not so perfect after all - a methodological study on patient-reported outcome measures in 2574 patients following percutaneous coronary intervention. Health Qual Life Outcomes. 2025 Apr 5;23(1):35. doi: 10.1186/s12955-025-02360-4. PMID 40188074
- [Derived] Hjertvikrem N, Brors G, Instenes I, Helmark C, Pettersen TR, Rotevatn S, Zwisler ADO, Norekval TM; CONCARDPCI Investigators. Use of health services and perceived need for information and follow-up after percutaneous coronary intervention. BMC Res Notes. 2024 Jan 5;17(1):20. doi: 10.1186/s13104-023-06662-y. PMID 38183067
- [Derived] Brors G, Dalen H, Allore H, Deaton C, Fridlund B, Norman CD, Palm P, Wentzel-Larsen T, Norekval TM. The association of electronic health literacy with behavioural and psychological coronary artery disease risk factors in patients after percutaneous coronary intervention: a 12-month follow-up study. Eur Heart J Digit Health. 2023 Feb 7;4(2):125-135. doi: 10.1093/ehjdh/ztad010. eCollection 2023 Mar. PMID 36974270
- [Derived] Ramstad KJ, Brors G, Pettersen TR, Deaton C, Palm P, Rotevatn S, Wentzel-Larsen T, Norekval TM. eHealth technology use and eHealth literacy after percutaneous coronary intervention. Eur J Cardiovasc Nurs. 2023 Jul 19;22(5):472-481. doi: 10.1093/eurjcn/zvac087. PMID 36190843
- [Derived] Brors G, Wentzel-Larsen T, Dalen H, Hansen TB, Norman CD, Wahl A, Norekval TM; CONCARD Investigators. Psychometric Properties of the Norwegian Version of the Electronic Health Literacy Scale (eHEALS) Among Patients After Percutaneous Coronary Intervention: Cross-Sectional Validation Study. J Med Internet Res. 2020 Jul 28;22(7):e17312. doi: 10.2196/17312. PMID 32720900
- [Derived] Norekval TM, Allore HG, Bendz B, Bjorvatn C, Borregaard B, Brors G, Deaton C, Falun N, Hadjistavropoulos H, Hansen TB, Igland S, Larsen AI, Palm P, Pettersen TR, Rasmussen TB, Schjott J, Sogaard R, Valaker I, Zwisler AD, Rotevatn S; CONCARD Investigators. Rethinking rehabilitation after percutaneous coronary intervention: a protocol of a multicentre cohort study on continuity of care, health literacy, adherence and costs at all care levels (the CONCARDPCI). BMJ Open. 2020 Feb 12;10(2):e031995. doi: 10.1136/bmjopen-2019-031995. PMID 32054625